CLINICAL TRIAL: NCT02378155
Title: Cerebral Oxygen Saturation Measurement During Cardioversion Because of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Cornelia Genbrugge, MD, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AF I
Record Dates: First submitted 2014-12-17; First posted 2015-03-04 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Electrical Cardioversion of Atrial Fibrillation; Pharmacological Cardioversion of Atrial Fibrillation
Keywords: cardioversion; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- electrical cardioversion (Other): Hemodynamic unstable patients with atrial fibrillation who are scheduled to undergo electrical reconversion to convert their irregular heart rhythm into a normal sinus rhythm. Cerebral tissue oxygen saturation is measured by means of SenSmart Model X-100, Nonin Medical.
  Interventions: Device: SenSmart Model X-100, Nonin Medical
- pharmacological cardioversion (Other): Patients who develop atrial fibrillation after cardiac surgery. Pharmacological treatment with amiodarone is started in order to convert their irregular heart rhythm into a normal sinus rhythm. Cerebral tissue oxygen saturation is measured by means of SenSmart Model X-100, Nonin Medical.
  Interventions: Device: SenSmart Model X-100, Nonin Medical

INTERVENTIONS:
Device: SenSmart Model X-100, Nonin Medical — Device to measure cerebral tissue oxygen saturation

SUMMARY:
Near infrared spectroscopy (NIRS) is a technique that measures regional cerebral oxygenation in a non-invasive manner. Through the use of near infrared light, the difference between oxygenated and deoxygenated hemoglobin can be measured. By applying the Lambert-Beer law, a numeric result can be calculated.

Since atrial fibrillation (AF) has been linked with an increased risk for the development of neurocognitive deficits, a longer period of AF might be associated with a higher risk for neurocognitive deficits.

It is hypothesized that there is an increase in the regional cerebral oxygen saturation (rSO2) of patients with paroxysmal or persistent AF after successful cardioversion.

DETAILED DESCRIPTION:
Written informed consent by the patient is asked before cardioversion and participation in the study. Patient anamnesis is assessed by standardized questionnaire.

Patients perform several standardised neurocognitive tests to obtain a general view on the neurocognitive status (auditory verbal learning test, mini-mental state examination, trail making A and B, digit-symbol coding and RAND 36 Health Survey).

Cerebral oxygenation is observed during cardioversion by means of the SenSmart Model X-100 (Nonin). Additional parameters (pulse oximetry, cardiac output, arterial blood pressure, 6-lead electrocardiography (ECG), left ventricular ejection fraction) are recorded. All measurements are performed non-invasively. Patients receive standard treatment following the clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years and able to give informed consent
* diagnosis of paroxysmal or persistent atrial fibrillation
* scheduled for electrical cardioversion or atrial fibrillation development in the first days after cardiac surgery followed by pharmacological treatment with amiodarone
* Dutch speaking

Exclusion Criteria:

* younger than 18 years or not able to give informed consent
* diagnosis of permanent atrial fibrillation
* atrial fibrillation with thrombus in left atrial appendage
* chronic obstructive pulmonary disease GOLD class 3 or 4
* airway manipulation during cardioversion
* pregnant women
* medical history of cerebrovascular accident or brain injury
* medical history of cardiopulmonary resuscitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Measure the cerebral saturation changes in response to electrical/pharmacological cardioversion | 6 months

SECONDARY OUTCOMES:
Measure the time for recuperation of cerebral saturation after a period of decreased cerebral saturation | 6 months
Relate the responses of cerebral saturation, regional saturation, pulse oximetry and blood pressure with each other | 6 months
Compare the changes in cerebral oxygen saturation with the left ventricular ejection fraction | 6 months
Perform neuropsychological tests before and after electrical/pharmacological cardioversion | 6 months
Compare the response of the cerebral/regional saturation with the effects on the neurocognitive status | 6 months
Compare the response of the pulse oximetry with the effects on the neurocognitive status | 6 months
Compare the response of the blood pressure with the effects on the neurocognitive status | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Genbrugge, MD, Principal Investigator — Hasselt University
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

REFERENCES:
- [Background] Pellicer A, Bravo Mdel C. Near-infrared spectroscopy: a methodology-focused review. Semin Fetal Neonatal Med. 2011 Feb;16(1):42-9. doi: 10.1016/j.siny.2010.05.003. Epub 2010 Jun 26. PMID 20580625
- [Background] Wutzler A, Nee J, Boldt LH, Kuhnle Y, Graser S, Schroder T, Haverkamp W, Storm C. Improvement of cerebral oxygen saturation after successful electrical cardioversion of atrial fibrillation. Europace. 2014 Feb;16(2):189-94. doi: 10.1093/europace/eut246. Epub 2013 Jul 31. PMID 23902651